CLINICAL TRIAL: NCT01640392
Title: Evaluating Locally Developed Homegrown HIV Prevention Interventions
Brief Title: MyLife MyStyle Evaluation Project
Acronym: MLMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Los Angeles County Department of Public Health (Other Government)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); In The Meantime Men's Group, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1 U01SP001573-01
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Unsafe Sex
Keywords: Gay men; African American males; Unprotected anal sex; HIV risk; behavioral intervention; group-level intervention
MeSH Terms: conditions — Unsafe Sex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIV prevention groups (Experimental): Participants randomly assigned to the MyLife Intervention arm receive three 1.5-hour HIV behavioral risk-reduction group sessions over a 1-3 week period.
  Interventions: Behavioral: MyLife MyStyle group-level intervention
- Wait-list control (No Intervention): Participants randomly assigned to the Wait-list Control arm receive the MyLife MyStyle group sessions once they have completed a 6-month follow-up assessment.

INTERVENTIONS:
Behavioral: MyLife MyStyle group-level intervention — Three 1.5-hour HIV behavioral risk-reduction group sessions conducted with up to 12 young African American/Black men (ages 18-29 years) over a 1-3 week period.
  Arms: HIV prevention groups

SUMMARY:
The purpose of the MyLife MyStyle Evaluation Project is to determine whether the MyLife MyStyle group-level intervention reduces HIV sexual-risk behaviors among 18- to 29-year-old African American men who have sex with men (MSM). Specifically, the project will test whether participants of the MyLife MyStyle program will report at least a 15% absolute decrease in frequency of unprotected anal sex with male partners at three and six months post-intervention compared with the wait-list control participants.

DETAILED DESCRIPTION:
In Los Angeles County, as well as nationally, the primary mode of HIV transmission for African American men is sexual contact with another man. According to national data from 45 states with name-based HIV surveillance in 2006, the majority of all new HIV infections among African American males were associated with sex with other men. The disproportionate impact of HIV in AAMSM in Los Angeles County is also observed in provisional HIV surveillance data. Between 2002 and 2004, AAMSM composed 16.3% of the new HIV diagnoses among males in Los Angeles County, with an average annual HIV diagnosis rate 2.0 and 2.5 times greater than the rates of new HIV diagnosis for White and Latino MSM, respectively. In addition to demonstrating the highest HIV prevalence and incidence estimates, AAMSM also had the highest proportion of previously unrecognized HIV infection (67%) compared with all other racial/ethnic groups. Given significant and continuing disparities in HIV infection among African Americans in the United States, and specifically among AAMSM, more intervention programs must be planned, implemented, and tested in order to reduce the heavy toll of HIV/AIDS in this population. Components of these intervention programs must be culturally competent and should include promotion of HIV counseling and testing to reduce the high prevalence of unrecognized HIV infection in AAMSM. Interventions should also take into consideration the many co-factors that may hinder AAMSM from addressing their HIV risk such as racism, poverty, stigma, and homophobia. The MyLife MyStyle Evaluation Project aims to implement and evaluate the efficacy of a "homegrown" group-level intervention to reduce HIV risk (unprotected anal sex with male partners) among young African American MSM in Los Angeles County, CA.

ELIGIBILITY:
Inclusion Criteria:

* Identify as African American or Black
* Identify as male
* Age 18 to 29 years
* Reside within Los Angeles County
* Self-reported anal sex with a male partner in the past 12 months
* Has not participated in an HIV prevention intervention in the past 3 months
* Able to complete ACASI and MyLife sessions in English

Exclusion Criteria:

* Identify as a transgender female
* Plan to move out of Los Angeles County before the end of their follow-up period (within 7 months)

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 528 (Actual)
Dates: Start 2012-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Reduced unprotected anal sex with male partners | up to 6 months following Intervention groups' third (final) session
  Proportion of intervention participants reporting any unprotected anal intercourse (either insertive or receptive) with male partners at six-month follow-up (and three months for short-term effects) compared with those in the wait-list control arm.

SECONDARY OUTCOMES:
Increased communication with partners | 3 months and 6 months following intervention groups' third (final) session
  Increase frequency of communication with partner(s) about safer sex, HIV status, STI status
Decrease unprotected sex because condom was not available | 3 months and 6 months following Intervention groups' third (final) session
  Proportion of intervention participants reporting episodes of unprotected anal sex when a condom is not available at six-month follow-up (and three months for short-term effects) compared with those in the wait-list control arm.
Decrease number of sexual partners | 3 months and 6 months following Intervention groups' third (final) session
  Number of sexual partners reported by intervention participants at six-month follow-up (and three months for short-term effects) compared with the number reported by the wait-list control participants.
Increase help-seeking behaviors for sexual health, e.g., STI testing, HIV testing, health screenings | 3 months and 6 months following Intervention groups' third (final) session
  Proportion of intervention participants reporting help-seeking behaviors for sexual health at six-month follow-up (and three months for short-term effects) compared with those in the wait-list control arm.

CONTACTS AND LOCATIONS:
Overall Officials: Trista Bingham, MPH, PhD, Principal Investigator — Los Angeles County Department of Public Health
Locations (1):
- In The Meantime Men's Group, Inc., Los Angeles, California, United States